CLINICAL TRIAL: NCT02845843
Title: MERS-CoV Infection tReated With A Combination of Lopinavir /Ritonavir and Interferon Beta-1b: a Multicenter, Placebo-controlled, Double-blind Randomized Trial
Brief Title: MERS-CoV Infection tReated With A Combination of Lopinavir /Ritonavir and Interferon Beta-1b
Acronym: MIRACLE
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: King Abdullah International Medical Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KingAbdullahIMRC
Record Dates: First submitted 2016-06-20; First posted 2016-07-27 (Estimated); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Middle East Respiratory Syndrome Coronavirus (MERS-CoV)
Keywords: Middle East Respiratory Syndrome Coronavirus; MERS-CoV; Clinical trial; Lopinavir; Ritonavir; Interferon beta
MeSH Terms: interventions — Ritonavir; Interferon beta-1b

STUDY DESIGN:
Intervention Model Description: This is a recursive two-stage group sequential multicenter placebo-controlled double-blind randomized controlled trial. The trial is initially designed to include 2 two-stage components. The first two-stage component is designed to adjust sample size and determine futility stopping, but not efficacy stopping (n=34). The second two-stage component is designed to determine efficacy stopping and possibly readjustment of sample size.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Combination of Lopinavir /Ritonavir and IntErferon Beta 1B (Experimental): Lopinavir /Ritonavir 400mg +100 mg / ml twice daily for 14 days and Interferon beta-1b 0.25 mg subcutaneous every alternate day for 14 days
  Interventions: Drug: Combination of Lopinavir /Ritonavir and Interferon beta-1b
- Placebo (Placebo Comparator): Same characteristics as Lopinavir /Ritonavir and Interferon beta-1b to maintain blinding
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Combination of Lopinavir /Ritonavir and Interferon beta-1b — Lopinavir /Ritonavir 400mg +100 mg / ml twice daily for 14 days and Interferon beta-1b 0.25 mg subcutaneous every alternate day for 14 days
  Arms: Combination of Lopinavir /Ritonavir and IntErferon Beta 1B
Drug: Placebo — Same characteristics as Lopinavir /Ritonavir and Interferon beta-1b to maintain blinding
  Arms: Placebo

SUMMARY:
This is a placebo-controlled clinical trial to assess the efficacy and safety of a combination of lopinavir/ritonavir and Interferon beta-1b in hospitalized patients with MERS.

DETAILED DESCRIPTION:
The aim of this study is to investigate the efficacy and safety of lopinavir /ritonavir and recombinant Interferon beta-1b combination given with optimal supportive care compared to placebo with optimal supportive care for patients with laboratory-confirmed MERS-CoV infection requiring hospital admission.

ELIGIBILITY:
Inclusion criteria at eligibility assessment

1. Adult (defined as ≥18 years of age);
2. Laboratory confirmation of MERS-CoV infection by reverse-transcription polymerase chain reaction (RT-PCR) from any diagnostic sampling source; and
3. New organ dysfunction that is judged to related to MERS including: hypoxia defined as requirement of supplemental oxygen to maintain oxygen saturations >90%, hypotension (systolic blood pressure<90 mmHg) or need for vasopressor/inotropic medication, renal impairment (increase of creatinine by 50% from baseline, glomerular filtration rate reduction by >25% from baseline or urine output of <0.5 ml/kg for 6 hours - Risk stage by RIFLE criteria), neurologic (reduction of Glasgow Coma Scale by 2 or more, i.e. 13 or lower of 15 points), thrombocytopenia (<150,000 platelets/mm3) or gastrointestinal symptoms that requires hospitalization (e.g. severe nausea, vomiting, diarrhea or/and abdominal pain).

Exclusion criteria at eligibility assessment

1. Suicidal ideation based on history (contraindication to interferon (IFN)-β1b);
2. Known allergy or hypersensitivity reaction to lopinavir/ritonavir or to recombinant IFN-β1b, including, but not limited to, toxic epidermal necrolysis, Stevens-Johnson syndrome, erythema multiforme, urticaria or angioedema;
3. Elevated alanine aminotransferase (ALT) >5 fold the upper limit in the hospital's laboratory;
4. Use of medications that are contraindicated with lopinavir/ritonavir and that cannot be replaced or stopped during the study period, such as CYP3A inhibitors;
5. Pregnancy - eligible and consenting female participants in childbearing age will be tested for pregnancy before enrollment in the study;
6. Known HIV infection, because of concerns about the development of resistance to lopinavir/ritonavir if used without combination with other anti-HIV drugs; or
7. Patient likely to be transferred to a non-participating hospital within 72 hours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2020-05 (Actual); Study Completion 2020-05 (Actual)

PRIMARY OUTCOMES:
90-day mortality | 90-day

SECONDARY OUTCOMES:
Organ support-free days (e.g., supplemental O2, ventilator, extracorporeal membrane oxygenation (ECMO), renal replacement and vasopressors) | 28 days
RT-PCR cycle threshold value in the lower respiratory samples | At randomization and every 3 days afterwards, until 2 consecutive samples are negative or reaching a maximum of 90 days
Sequential organ failure assessment (SOFA) scores | Days 0, 3, 7, 14, 21 and 28
ICU-free days | Number of days in which patients are not being cared for in the ICU during the first 28 days after enrollment
Length of stay in hospital | Up to one year from enrollment
Number of Patients with Adverse drug reactions related to the treatment | From enrollment to 28 day
Karnofsky Performance Scale | 90-day
ICU mortality | Up to one year from enrollment
Hospital mortality | Up to one year from enrollment
28-day mortality | 28-day

CONTACTS AND LOCATIONS:
Locations (2):
- Saudi Arabia (2):
  - Intensive Care Unit, King Abdulaziz Medical City, National Guard Health Affairs, Riyadh
  - King Abdullah International Medical Research Center, Riyadh

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Arabi YM, Asiri AY, Assiri AM, Abdullah ML, Aljami HA, Balkhy HH, Al Jeraisy M, Mandourah Y, AlJohani S, Al Harbi S, Jokhdar HAA, Deeb AM, Memish ZA, Jose J, Ghazal S, Al Faraj S, Al Mekhlafi GA, Sherbeeni NM, Elzein FE, Hayden FG, Fowler RA, AlMutairi BM, Al-Dawood A, Alharbi NK. Heterogeneity of treatment effect of interferon-beta1b and lopinavir-ritonavir in patients with Middle East respiratory syndrome by cytokine levels. Sci Rep. 2022 Oct 28;12(1):18186. doi: 10.1038/s41598-022-22742-8. PMID 36307462
- [Derived] Arabi YM, Asiri AY, Assiri AM, Balkhy HH, Al Bshabshe A, Al Jeraisy M, Mandourah Y, Azzam MHA, Bin Eshaq AM, Al Johani S, Al Harbi S, Jokhdar HAA, Deeb AM, Memish ZA, Jose J, Ghazal S, Al Faraj S, Al Mekhlafi GA, Sherbeeni NM, Elzein FE, Al-Hameed F, Al Saedi A, Alharbi NK, Fowler RA, Hayden FG, Al-Dawood A, Abdelzaher M, Bajhmom W, AlMutairi BM, Hussein MA, Alothman A; Saudi Critical Care Trials Group. Interferon Beta-1b and Lopinavir-Ritonavir for Middle East Respiratory Syndrome. N Engl J Med. 2020 Oct 22;383(17):1645-1656. doi: 10.1056/NEJMoa2015294. Epub 2020 Oct 7. PMID 33026741
- [Derived] Arabi YM, Asiri AY, Assiri AM, Aziz Jokhdar HA, Alothman A, Balkhy HH, AlJohani S, Al Harbi S, Kojan S, Al Jeraisy M, Deeb AM, Memish ZA, Ghazal S, Al Faraj S, Al-Hameed F, AlSaedi A, Mandourah Y, Al Mekhlafi GA, Sherbeeni NM, Elzein FE, Almotairi A, Al Bshabshe A, Kharaba A, Jose J, Al Harthy A, Al Sulaiman M, Mady A, Fowler RA, Hayden FG, Al-Dawood A, Abdelzaher M, Bajhmom W, Hussein MA; and the Saudi Critical Care Trials group. Treatment of Middle East respiratory syndrome with a combination of lopinavir/ritonavir and interferon-beta1b (MIRACLE trial): statistical analysis plan for a recursive two-stage group sequential randomized controlled trial. Trials. 2020 Jan 3;21(1):8. doi: 10.1186/s13063-019-3846-x. PMID 31900204
- [Derived] Arabi YM, Alothman A, Balkhy HH, Al-Dawood A, AlJohani S, Al Harbi S, Kojan S, Al Jeraisy M, Deeb AM, Assiri AM, Al-Hameed F, AlSaedi A, Mandourah Y, Almekhlafi GA, Sherbeeni NM, Elzein FE, Memon J, Taha Y, Almotairi A, Maghrabi KA, Qushmaq I, Al Bshabshe A, Kharaba A, Shalhoub S, Jose J, Fowler RA, Hayden FG, Hussein MA; And the MIRACLE trial group. Treatment of Middle East Respiratory Syndrome with a combination of lopinavir-ritonavir and interferon-beta1b (MIRACLE trial): study protocol for a randomized controlled trial. Trials. 2018 Jan 30;19(1):81. doi: 10.1186/s13063-017-2427-0. PMID 29382391